CLINICAL TRIAL: NCT02985606
Title: How Does Altering the Timing of Pre-exercise Low-dose Caffeine Ingestion Affect Endurance Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 181739/02
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Caffeine -60 (Active Comparator): Caffeine at 60 minutes prior to time trial
  Interventions: Other: Caffeine powder -60; Other: Placebo powder -30; Other: Placebo powder 0
- Caffeine -30 (Active Comparator): Caffeine at 30 minutes prior to time trial
  Interventions: Other: Caffeine powder -30; Other: Placebo powder -60; Other: Placebo powder 0
- Caffeine 0 (Active Comparator): Caffeine immediately prior to time trial
  Interventions: Other: Caffeine powder 0; Other: Placebo powder -60; Other: Placebo powder -30
- Placebo (Placebo Comparator): Placebo drink at all time points
  Interventions: Other: Placebo powder -60; Other: Placebo powder -30; Other: Placebo powder 0

INTERVENTIONS:
Other: Caffeine powder -60
  Arms: Caffeine -60
Other: Caffeine powder -30
  Arms: Caffeine -30
Other: Caffeine powder 0
  Arms: Caffeine 0
Other: Placebo powder -60
  Arms: Caffeine -30; Caffeine 0; Placebo
Other: Placebo powder -30
  Arms: Caffeine -60; Caffeine 0; Placebo
Other: Placebo powder 0
  Arms: Caffeine -30; Caffeine -60; Placebo

SUMMARY:
Investigate how manipulating the time between caffeine ingestion and exercise may alter exercise performance and cognition

ELIGIBILITY:
Inclusion Criteria:

* vo2max > 55 ml/kg/min
* females on contraceptive pill

Exclusion Criteria:

* recent skeletal muscle injury
* cardiovascular injury
* metabolic disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06-30 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Work done in kilojoules (kJ) during a 15 minute time trial on a cycle ergometer | 15 minutes

SECONDARY OUTCOMES:
Whole body fuel substrate utilisation measured using indirect calorimetry | 10 minutes
Change in plasma caffeine concentration and metabolites | 2 hours 45 minutes
Change in cognitive function measured using stroop test | 2 hours 45 minutes
Collection of saliva for genotyping of CYP1A2 | 30 mintes

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Health Sciences, Exeter, Devon, United Kingdom

REFERENCES:
- [Derived] Davenport AD, Jameson TSO, Kilroe SP, Monteyne AJ, Pavis GF, Wall BT, Dirks ML, Alamdari N, Mikus CR, Stephens FB. A Randomised, Placebo-Controlled, Crossover Study Investigating the Optimal Timing of a Caffeine-Containing Supplement for Exercise Performance. Sports Med Open. 2020 Mar 30;6(1):17. doi: 10.1186/s40798-020-00246-x. PMID 32232597